CLINICAL TRIAL: NCT00373698
Title: Reengineering Systems for the Primary Care Treatment of PTSD
Brief Title: Re-Engineering Systems for the Primary Care Treatment for PTSD
Acronym: RESPECT-PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAC 06-073
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-06

CONDITIONS: Stress Disorders, Posttraumatic; Depression
Keywords: Stress Disorders, Posttraumatic; Delivery of Health Care, Integrated; Primary Health Care; Veterans; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three Component Model (Experimental): Three Component Model of Collaborative Care: Patients randomized to 3CM will receive telephone care management along with usual care by VA clinicians.
  Interventions: Behavioral: Three Component Model of Collaborative Care
- Usual Care (No Intervention): Patients randomized to "Usual Care" will receive care as usual by VA clinicians.

INTERVENTIONS:
Behavioral: Three Component Model of Collaborative Care — Patients randomized to 3CM will receive telephone care management along with usual care by VA clinicians.
  Arms: Three Component Model

SUMMARY:
The study is an evaluation of a systemic intervention to enhance the delivery of care according to practice guidelines for posttraumatic stress disorder (PTSD). The immediate objectives are to (1) implement three component model (3CM) in VA primary care clinics; and (2) evaluate the effects of 3CM on clinician behavior and patient outcomes. The long-term objectives are to generate information to support implementation research on the RESPECT model for treating PTSD in primary care and ultimately, the implementation of the model in VHA to provide care to veterans with PTSD.

DETAILED DESCRIPTION:
3CM consists of (1) a prepared practice, (2) care management, and (3) enhanced mental health support. A prepared practice refers to education for primary care clinicians and office staff about practice guidelines and evidence-based care, the skills needed for use of assessment measures, and the use of communication forms and routines. The education plan consists of predisposing activities, including active teaching and learning, and enabling and reinforcing activities in order to help clinicians use newly acquired skills and to reinforce the continued use of these skills in practice. Care management is accomplished by telephone, usually by a centrally located care manager during acute phase treatment and follow up to answer patient questions, promote adherence to the clinician's management plan, and help patients overcome barriers to adherence. Enhanced mental health support is provided by a psychiatrist who supervises care managers by telephone, provides informal consultation to primary care clinicians, and helps to increase the quantity or quality of mental health referral resources.

ELIGIBILITY:
Inclusion Criteria:

* Military Veterans in Primary Care Clinics who meet diagnostic criteria for PTSD in one of the 5 sites in Texas where this study is being conducted.
* Must have regular access to a telephone and speak English.

Exclusion Criteria:

* Cognitive impairment
* A history of psychosis or mania
* Prominent current suicidal ideation
* Current substance dependence
* Current engagement in mental health treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula P Schnurr, PhD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (4):
- United States (4):
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

REFERENCES:
- [Result] Schnurr PP, Friedman MJ, Oxman TE, Dietrich AJ, Smith MW, Shiner B, Forshay E, Gui J, Thurston V. RESPECT-PTSD: re-engineering systems for the primary care treatment of PTSD, a randomized controlled trial. J Gen Intern Med. 2013 Jan;28(1):32-40. doi: 10.1007/s11606-012-2166-6. Epub 2012 Aug 3. PMID 22865017

RESULTS

PARTICIPANT FLOW:
Groups:
- Three Component Model of Collaborative Care and Usual Care: Participants randomized to this arm received the Three Component Model of Collaborative Care (3CM) as well as usual care. 3CM model consists of 1) education and tools for primary care clinicians and staff including content regarding PTSD; 2) telephone care management by a centrally located care manager (the purpose of the calls was to identify barriers to adherance with the primary care provider's plan, aid participant to overcome them, and measure treatment response. Calls occurred 1, 4, and 8 weeks after the initial visit and then every 4 weeks for 6 months or until a participant acheived 30% reduction in PTSD symptoms as measure by the PCL); 3) support from a psychiatrist who supervises care managers by telephone, provides consultation to primary care clinicians, and facilitates mental health referral. Participant's "Usual Care" is at the VA provider's discretion and could include referral to mental health specialty care.specialty care.
- Usual Care: Participants randomized to "Usual Care" received care at the VA provider's discretion and could include referral to mental health specialty care.
Period: Overall Study
Arm/Group | Three Component Model of Collaborative Care and Usual Care | Usual Care
Started | 96 | 99
Completed | 85 | 99
Not Completed | 11 | 0

BASELINE CHARACTERISTICS:
Population: To be included, subjects had to meet diagnostic criteria for PTSD, have regular access to a telephone, and speak English. Exclusion criteria were cognitive impairment, history of psychosis or mania, prominent current suicidal ideation, current substance dependence, and current engagement in mental health treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Three Component Model | Usual Care | Total
Number analyzed (Participants) | 96 | 99 | 195
Age, Customized [Mean (Full Range); unit: years]
  Age, >=18 | 46.1 [NA to NA] — 43.1-49.1 (95% confidence interval) | 44.4 [NA to NA] — 41.3-47.5 (95% confidence interval) | NA [NA to NA] — The data are locked and the total can not be calculated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 89 | 89 | 178
Region of Enrollment [Number; unit: participants]
  United States | 96 | 99 | 195
PTSD symptom severity (used Posttraumatic Diagnostic Scale (PDS)) [Mean (Standard Deviation); unit: units on a scale] — The PDS yields a total severity score (ranging from 0 to 51, where 0 is the best and 51 is the worst) that largely reflects the frequency of the 17 symptoms of PTSD. 17 symptoms of PTSD are rated individually on a scale from 0 to 3, with 3 being the highest. Total severity score is calculated by adding the number from each individual symptom. A PDS Profile Report also provides a preliminary determination of DSM-IV PTSD diagnostic status, a count of the number of symptoms endorsed, a rating of symptom severity, and a rating of the level of impairment of functioning.
  units on a scale | 33.2 (8.3) | 34.0 (9.7) | NA (NA) — The data are locked and can not be calculated
Depression (Hopkins Symptom Checklist-20) [Mean (Standard Deviation); unit: units on a scale] — Depression severity (ranging 0-4) was measured with the Hopkins Symptom Checklist-20. This self-assessment measure consists of 20 questions with possible scores ranging from 0 to 4, with higher scores indicating worse symptoms. Means and the standard deviations of the 20 questions are presented with higher scores indicating worse depression.
  units on a scale | 1.98 (0.69) | 2.06 (0.78) | NA (NA) — The data are locked and can not be calculated
SF-36 Mental Component [Mean (Standard Deviation); unit: units on a scale] — SF-36 Mental Component is measured as part of SF-36 Health Survey. Scores can range from 0 (poorest possible health ) to 100 (highest possible health).
  units on a scale | 33.8 (8.8) | 32.7 (8.1) | NA (NA) — The data are locked and can not be calculated.
SF-36 Physical Component [Mean (Standard Deviation); unit: units on a scale] — SF-36 Physical Component is measured as part of SF-36 Health Survey. Scores can range from 0 (poorest possible health ) to 100 (highest possible health).
  units on a scale | 42.2 (13.0) | 43.4 (12.6) | NA (NA) — The data are locked and can not be calculated.

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity
Description: PTSD Symptom Severity was measured using the Postraumatic Diagnostic Scale (PDS)
Time Frame: 3 and 6 months after initial assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm1/Three Component Model of Care Collaborative Care: Three Component Model of Collaborative Care: Patients randomized to 3CM will receive telephone care management along with usual care by VA clinicians.
- Arm 2/Usual Care: Patients randomized to "Usual Care" will receive care as usual by VA clinicians.
Arm/Group | Arm1/Three Component Model of Care Collaborative Care | Arm 2/Usual Care
Number analyzed (Participants) | 96 | 99
units on a scale
  3 months after initial assessment | 31.4 (10.2) | 31.5 (10.3)
  6 months after initial assessment | 30.2 (10.3) | 29.9 (10.8)

2. Secondary Outcome: Depression
Description: Measure using the Hopkins Symptom Checklist-20
Time Frame: 3 and 6 months after initial assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm1/Three Component Model of Care Collaborative Care | Arm 2/Usual Care
Number analyzed (Participants) | 96 | 99
units on a scale
  3 months after initial assessment | 1.8 (0.8) | 1.84 (0.82)
  6 months after initial assessment | 1.81 (0.84) | 1.83 (0.90)

3. Secondary Outcome: SF-36 Mental Component
Time Frame: 3 and 6 months after initial assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm1/Three Component Model of Care Collaborative Care | Arm 2/Usual Care
Number analyzed (Participants) | 96 | 99
units on a scale
  Mental Component-3 months after initial assessment | 33.9 (8.3) | 33.8 (8.1)
  Mental Component-6 months after initial assessment | 33.7 (9.4) | 33.4 (8.1)

4. Secondary Outcome: SF-36 Physical Component
Time Frame: 3 and 6 months after initial assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Three Component Model | Usual Care
Number analyzed (Participants) | 96 | 99
units on a scale
  Physical Component-3 months after initial assessme | 43.8 (13.1) | 43.7 (12.2)
  Physical Component-6 monthsafter initial assessmen | 44.4 (12.6) | 44.8 (11.8)

ADVERSE EVENTS:
Arm/Group | Three Component Model | Usual Care
Serious Adverse Events (participants affected / at risk) | 5/96 | 4/99
Other Adverse Events (participants affected / at risk) | 0/96 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Three Component Model (N=96) | Usual Care (N=99)
hospitalization (Surgical and medical procedures) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes